CLINICAL TRIAL: NCT02757417
Title: A Randomized Trial Comparing Intaoperative Intravenous Sodium Fluorescein to Pre-Operative Oral Phenazopyridine For Evaluation of Ureteral Patency
Brief Title: Intravenous Sodium Fluorescein Versus Oral Phenazopyridine for Ureteral Patency
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Megan Billow (Unknown); Graham Chapman (Unknown); Sangeeta Mahajan (Unknown); Alex Soriano (Unknown); Sherif El-Nashar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UHcaseMC1
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Ureteral Injury
MeSH Terms: interventions — Fluorescein; Phenazopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Fluorescein (Active Comparator): Patients will receive an intravenous dose of 0.25 mL of 10% (500 mg, 5 mL) sodium fluorescein at the time of cystoscope insertion, for a total dose of 25 mg. Cystoscopy will be performed in the standard fashion during the course of the operation.
  Interventions: Drug: sodium fluorescein
- oral phenazopyridine (Active Comparator): Patients randomized to the phenazopyridine arm will be given a 200 mg pill with a sip of water in the pre-operative area 1 hour before their scheduled procedure. Cystoscopy will be performed in the standard fashion during the course of the operation.
  Interventions: Drug: phenazopyridine

INTERVENTIONS:
Drug: sodium fluorescein
  Arms: Sodium Fluorescein
Drug: phenazopyridine
  Arms: oral phenazopyridine

SUMMARY:
To determine the safety profile of sodium fluorescein in women undergoing cystoscopy during gynecologic surgery. To determine if either oral phenazopyridine or sodium fluorescein result in shorter cystoscopy times.

ELIGIBILITY:
Inclusion Criteria:

* - Patients must be 18 years or older as well as willing and able to provide informed consent
* Patients undergoing a scheduled gynecologic procedure with cystoscopy

Exclusion Criteria:

* - Patients are younger than 18 years
* Patients are unable or unwilling to provide informed consent
* Patients with a history of an allergic reaction to sodium fluorescein or phenazopyridine
* Patients with a history of renal insufficiency
* Patients with a history of liver disease
* Patients with a history of sickle cell disease
* Patients with a history of glucose-6-phosphate dehydrogenase deficiency
* Patients with a history of chronic obstructive pulmonary disease or currently being treated for asthma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
differences in time that elapses between starting cystoscopy and identifying both ureteral jets between treatment groups | 12 months

SECONDARY OUTCOMES:
number of participants with intra-operative and immediate and post-operative treatment-related adverse events as assessed by CTCAE v4.0 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided